CLINICAL TRIAL: NCT01453114
Title: Cognitive-Behavioral Therapy in Women Discontinuing Antidepressant for Pregnancy
Brief Title: Cognitive-Behavioral Therapy (CBT) in Women Discontinuing Antidepressant for Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Lee S. Cohen, MD, Director of the Perinatal and Reproductive Psychiatry Clinical Research Program, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2008P002161
Record Dates: First submitted 2011-10-12; First posted 2011-10-17 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2015-04

CONDITIONS: Depression; Postpartum Depression; Antenatal Depression
Keywords: Cognitive Behavioral Therapy; CBT; relapse; postpartum depression; depression recurrence; depression relapse
MeSH Terms: conditions — Depression; Depression, Postpartum; Recurrence | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Psychotherapy (Experimental): Cognitive Behavioral Therapy
  Interventions: Behavioral: Cognitive Behavioral Therapy

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy — CBT is administered for 12 sessions over the period of 16 weeks, followed by optional monthly sessions.
  Other Names: CBT

SUMMARY:
The overarching goal of this study is to adapt a cognitive behavioral prevention of recurrence treatment (CBT-PR) for women with a history of recurrent major depressive disorder who decide to discontinue their maintenance anti-depressant (AD) treatment for pregnancy.

DETAILED DESCRIPTION:
The current study is a small year-long pilot to collect data for a planned larger, randomized control trial in the future. The current protocol focuses on modifying a Cognitive-Behavioral Therapy (CBT) recurrence prevention protocol for the study population, finalizing a therapist training manual, finalizing therapist adherence and competence scales, and fine tuning research procedures for recruitment and retention of subjects. This phase will involve enrolling 20 subjects in order to have at least 12 subjects receive CBT treatment for 12 weeks with assessments conducted bimonthly. The subjects will have the option of having additional monthly "booster" CBT sessions. Independent Assessments by HRC-approved study staff and interviews with study psychiatrists will occur at 16 weeks, 24 weeks, 36 weeks, and 1 year after study initiation. Participants will be offered the opportunity to speak with a study psychiatrist at every visit.

The primary outcome measure is rate of recurrence and/or re-initiation of antidepressant treatment up to 12 months post-randomization. The study end point of procedures is 12 weeks after baseline; the study end point for follow-up assessments is one year after treatment.

At the point of enrollment, subjects will have reviewed risks and benefits of perinatal depression treatment in a consultation with a non-study psychiatrist in the MGH Center for Women's Mental Health (CWMH) program and in collaboration with the subject's primary psychiatrist, and decided to discontinue AD treatment.

The potential subject will then undergo a preliminary phone screening with a CWMH research coordinator where basic eligibility criteria are reviewed. If the potential subject is interested, she will be scheduled for a baseline study visit conducted by the PIs or another study clinician. After an explanation of study procedures, written, informed consent will be obtained. This will occur prior to execution of any study assessments or procedures.

After consent is obtained, the clinician will conduct a structured clinical interview using the MINI and HRC-approved study staff will complete study assessments. If the potential subject continues to be interested in participating in the study and remains eligible, she will meet with a study psychiatrist who will instruct her on how to begin the taper of her antidepressant, if she has not already started to taper. The subject will then meet with the clinician who will administer the CBT treatment for the first session

After the 12 weeks have passed, subjects will be asked to complete assessments at 16 weeks, 24 weeks, 36 weeks, and 1 year after beginning the study, and will be able to choose to continue monthly booster sessions of CBT-PR. Subjects will also be offered the opportunity to meet with study psychiatrists every booster session. Visits with the study psychiatrist will be arranged at the discretion of the study psychologist and/or upon participant request. An optional qualitative interview will be conducted by study staff after completion of the acute treatment phase in order to obtain feedback on the intervention.

Participants who experience a relapse of depressive symptoms during study participation will have the option of remaining in the study and continuing to receive CBT treatment regardless of decisions regarding antidepressant treatment. Additionally, the investigators will ask patients who experience a relapse to complete a questionnaire regarding the course of relapse and their treatment decisions at one year after study enrollment. This questionnaire can be completed over the phone or at home and returned by mail.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will include women 18 years and older who are either planning pregnancy or already pregnant and meet the following criteria:
* Currently meet criteria for stable remission from depression (defined as a baseline score of ≤ 9 on the Hamilton Rating Scale for Depression (HRSD) and documented clinical remission for a minimum of six months prior to randomization)
* Current or recent treatment with an antidepressant (stable dosage for at least the last four weeks)
* Have a history of a major depressive episode
* Decide to discontinue antidepressant medication for pregnancy
* Currently receive ongoing psychiatric care provided by a physician outside the MGH Center for Women's Mental Health, and written, informed consent.

Exclusion Criteria:

* Significant risk for self-harm or harm to others
* Psychotic symptoms
* Meeting criteria for a primary SCID-I/P diagnosis of schizophrenia, bipolar disorder, an active eating disorder, dementia, delirium, or other cognitive disorder
* Presence of an active substance and/or alcohol abuse disorder within six months prior to screening visit
* Current use of mood stabilizers, antipsychotics or antiepileptics
* Have received cognitive-behavioral or interpersonal therapy within the last year
* Diagnosed with a medical disorder that has a known association with depressive symptoms (e. g. thyroid disorder).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2008-11; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Relapse | Within a year of study entry
  MDE diagnosed using the mood module of the Mini-International Neuropsychiatric Interview (MINI)

SECONDARY OUTCOMES:
Depression severity | throughout the 52 weeks of the study
  Depression severity is determined using the Montgomery-Asberg Depression Rating Scale (MADRS).

CONTACTS AND LOCATIONS:
Overall Officials: Lee S Cohen, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States